CLINICAL TRIAL: NCT07196462
Title: Precision Brain Stimulation to Reduce Cannabis Craving in Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Heather Burrell Ward, Principle Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 250955
Record Dates: First submitted 2025-09-13; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use; SCHIZOPHRENIA; Psychosis; rTMS
Keywords: cannabis use; schizophrenia; rTMS; brain stimulation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Precision Brain Stimulation for Cannabis Users with Schizophrenia (Experimental): Participants with schizophrenia who use cannabis.
  Interventions: Device: 3 Minute iTBS to the L DLPFC; Device: One-Minute, Personalized, DMN Targeted CTBS
- Precision Brain Stimulation for Cannabis Users with Healthy Controls (Active Comparator): Healthy controls who use cannabis.
  Interventions: Device: 3 Minute iTBS to the L DLPFC; Device: One-Minute, Personalized, DMN Targeted CTBS

INTERVENTIONS:
Device: 3 Minute iTBS to the L DLPFC — Five daily sessions of TMS (iTBS) to the L DLPFC target.
Device: One-Minute, Personalized, DMN Targeted CTBS — Personalized, DMN Targeted CTBS to the DMN for one minute, five daily sessions.

SUMMARY:
The central hypothesis is this: Brain circuits most relevant to cannabis use in schizophrenia are distinct from pathways identified in healthy controls who use cannabis. This study seeks to provide evidence that targeted stimulation of the DMN leads to both altered network activity and a concomitant behavioral change in cue-induced craving and cognitive performance in individuals with schizophrenia and schizoaffective disorder, while targeted stimulation of the L DLPFC leads to these changes in healthy controls who use cannabis. This study will test a model that integrates brain network pathophysiology and cognition to 1) explain the prevalence of cannabis use in schizophrenia and 2) identify a target for engagement in schizophrenia. This study seeks to establish a neuroscientific framework to guide future treatment-oriented studies aimed at reducing craving and improving cognitive performance in individuals with schizophrenia and schizoaffective disorder.

This is a study of the effect of 2 rTMS interventions on functional connectivity and craving in individuals with schizophrenia or schizoaffective disorder and healthy controls who use cannabis.

Aim 1: Target Engagement: Determine if rTMS manipulates functional connectivity of each target (DMN, L DLPFC) (n=100).

Aim 2: Clinical Efficacy: Determine if rTMS affects cue-induced craving and if craving change correlates with change in functional connectivity (n=100).

As an exploratory analysis, the factors that explain individual variance in rTMS-induced connectivity change will also be explored.

DETAILED DESCRIPTION:
Cannabis use is highly prevalent in schizophrenia and has devastating consequences but no current treatments. Psychotic disorders such as schizophrenia are disabling, lifelong illnesses that afflict over three million people in the US. Cannabis is the second-most commonly used substance by people with schizophrenia (SZ) after tobacco. Up to 43% of people with SZ meet criteria for cannabis use disorder (CUD), a rate 15 times that in the general population of 3%. Recent evidence suggests cannabis use and SZ have bidirectional causal relationships. Co-occurring SZ with CUD has a significantly worse prognosis than SZ alone, as CUD is associated with symptom exacerbation, risk of psychotic relapse, treatment nonadherence, and poorer overall functioning. Cannabis use is a frequent cause of medication nonadherence, psychotic decompensation, and psychiatric hospitalization. Cannabis use in adolescence commonly occurs prior to the onset of psychosis, and there is growing evidence that cannabis may cause schizophrenia in vulnerable individuals. Recent evidence shows that cannabis use triggers brain changes linked to psychosis. However, the underlying pathophysiology of SZ with CUD remains unknown, and there are no approved treatments for SZ with CUD, leaving patients and their families struggling to stop their cannabis use without any effective treatments.

Cannabis Use in Schizophrenia is Based in Brain Network Pathology. Despite the magnitude of cannabis use and its devastating consequences, there are no approved treatments for cannabis use in any population. This study team seeks to investigate if this vulnerability to cannabis use in schizophrenia is based in brain pathology. The human brain is organized into networks of connected regions. In cannabis users, a region of these networks is chronically hyperconnected, but cannabis use transiently corrects this network pathology. This suggests cannabis users are using cannabis to self-medicate a network pathology problem. Function of brain networks can be measured in the MRI scanner.

This study seeks to use functional connectivity as a measure of neural function. The human brain has evolved to perform different behaviors under different sets of conditions and as such must flexibly combine the functional processing capabilities of disparate neuroanatomical regions. Collections of structurally interconnected brain areas must interact dynamically to process a large and ever-changing set of inputs in the ultimate attempt to generate an appropriate behavioral output. Functional networks can therefore be defined as the collection of interconnected brain areas that interact to perform these circumscribed functions.

To identify the critical nodes involved in these different functional networks, much of the work in the field of functional neuroimaging has used the fMRI blood-oxygen-level-dependent (BOLD) signal as a marker of cerebral perfusion, which in turn is known to reflect cerebral activity. fMRI BOLD activation patterns have revealed network nodes that are involved in such cognitive functions as attention working memory, language, and others.

In the resting state--while a participant is asked simply to look straight without performing a specific task in the MRI--analyses of the time-course of BOLD activation have revealed that activity patterns of several of these cerebral nodes exhibit coordinated fluctuations. As such, the activity patterns between particular nodes appear to be highly correlated in time while others seem relatively independent of one another. Taken together, these coordinated nodes can be thought of as a coupled functional network. The correlations between the activity patterns of cerebral nodes are termed "functional connectivity."

DMN Hyperconnectivity is associated with cannabis use and is improved by cannabis administration. In healthy cannabis users, parietal default mode network (DMN) hyperconnectivity has been observed during rest and task conditions. Moreover, the parietal DMN activates to cannabis cues, and cannabis administration reduces parietal DMN connectivity.

The relationship will also be observed in psychosis: in a large sample of individuals with psychosis (Prelim Data #1, n= 596), higher DMN connectivity was related to more lifetime cannabis use. Higher DMN connectivity was also associated with higher craving in SZ (Prelim Data #2, r=0.49, p=.0097).

DMN hyperconnectivity is a well-established observation in SZ. Critically, the only study of cannabis administration among SZ with CUD showed that both cannabis and THC normalized DMN hyperconnectivity to the level of healthy controls (Whitfield-Gabrieli et al. 2018). These convergent data suggest that parietal DMN hyperconnectivity in SZ may be further exacerbated by cannabis use, suggesting the parietal DMN may be a prime target for intervention.

5) rTMS is an FDA-Approved Treatment for Substance Use that Can Selectively Target Brain Network Pathology TMS, (Transcranial Magnetic Stimulation) is a non-invasive, easily transportable, and relatively inexpensive procedure that utilizes magnetic fields to create electric currents in discrete brain regions. TMS is based on Faraday's principle of electromagnetic induction and features application of rapidly changing magnetic field pulses to the scalp via a copper wire coil connected to a magnetic stimulator. These brief pulsed magnetic fields painlessly pass through the skull and create electric currents in discrete brain regions of sufficient magnitude to depolarize neurons. Applied in single pulses (single-pulse TMS) appropriately delivered in time and space, the currents induced in the brain can be of sufficient magnitude to depolarize a population of neurons. When applied to the motor cortex, this depolarization results in a series of descending (direct and indirect) corticospinal waves that can sum-up at the spinal segmental level, depolarize alpha motor neurons and lead to the contraction of contralateral muscles. This can be measured, for example, as motor evoked potentials (MEPs) using electromyography (EMG). Applied to any cortical region, TMS evokes a local field potential that can be recorded with EEG, or other brain imaging techniques, and reveals a measure of cortical reactivity to TMS. TMS intensity can be parametrically varied in its intensity thus allowing the establishment of a dose-response curve and providing insights into cortical excitability.

Trains of repeated TMS pulses (rTMS) at various stimulation frequencies and patterns can induce a lasting modification of activity in the targeted brain region which can outlast the effects of the stimulation itself. Such lasting changes presumably represent alterations in plasticity mechanisms. Therefore, rTMS can be used with repeated pulses to facilitate activity in a region of the brain or suppress activity in a region of the brain.

When international safety guidelines are followed, rTMS is a safe and well-tolerated intervention for people with and without psychiatric illness. rTMS is currently an FDA-approved treatment for major depressive disorder, obsessive-compulsive disorder, and smoking cessation. FDA-approved treatment for major depressive disorder generally involves 20-30 daily sessions of rTMS delivered to the left dorsolateral prefrontal cortex (L DLPFC). However, the FDA recently cleared the SAINT protocol for depression, which involves a total of 50 sessions over 5 days (10 sessions/day). FDA-approved treatment for smoking cessation involves treatment to the L and R DLPFC and has been shown to significantly reduce cigarette consumption and craving in smokers without psychiatric illness.

rTMS is a Safe and Effective Treatment for People with Schizophrenia. rTMS has been studied in thousands of people with schizophrenia for a number of different indications, for example auditory verbal hallucinations (systematic review of n = 960 participants), negative symptoms (systematic review, n = 2633 participants), cognitive deficits (systematic review, n = 351 participants) and nicotine dependence. In a meta-analysis of the safety of rTMS in schizophrenia conducted by the PI, it was found that the prevalence of side effects from rTMS for individuals with schizophrenia was at or below the prevalence in the general population. People with schizophrenia were NOT at higher risk for worsening of psychiatric symptoms or seizure.

Notably, rTMS is approved for suppression of treatment-refractory auditory hallucinations in schizophrenia by the National Institutes of Mental Health (NIMH). Additionally, a systematic review of 524 individuals with schizophrenia who received intermittent theta burst stimulation (i.e. excitatory theta burst TMS), they noted, "Overall iTBS was well tolerated in patients with schizophrenia". There were no significant differences observed in adverse events between active and sham iTBS, and no seizures were reported. The Safety of TMS Consensus Group recommended, "available data indicate no additional risks of major AEs [adverse events] in specific patient populations [including schizophrenia] so this is not a concern that needs to be taken into account, at least with the protocols of intervention considered" . No seizures were observed in any of these systematic reviews.

rTMS is a Safe and Effective Treatment for Substance Use Disorders, Including Cannabis User. TMS is FDA-approved for treatment of nicotine use disorder and has been tested in thousands of individuals with substance use disorders (Mehta et al. 2023). rTMS for cannabis use disorder has been studied in multiple studies in both the general population and in schizophrenia without any safety concerns. In schizophrenia, 20 sessions of rTMS applied to the DLPFC led to reductions in cannabis use and improvement in cognitive performance.

Past studies by this research group have conducted rTMS studies showing that Default Mode Network-targeted cTBS reduces DMN connectivity. In Prelim Data #3, individuals with SZ received single sessions of Default Mode Network-targeted cTBS (active and sham) with MRI immediately before and after rTMS. Past studies have observed that Default Mode Network-targeted cTBS reduced DMN connectivity compared to sham rTMS (p=.0028, Figure 2). Previously, this research team has also conducted rTMS studies showing that Default Mode Network-targeted cTBS in SZ reduces craving, while Conventional DLPFC-targeted iTBS does not (Prelim Data #4). As pilot data for the proposed study, individuals with SZ underwent 5 daily sessions of 1) Default Mode Network-targeted cTBS and 2) Conventional DLFPC-targeted iTBS in a crossover design with MRI and craving assessment before and after each rTMS week. It was observed that only Default Mode Network-targeted cTBS significantly reduced craving in SZ (n=7, p<.05).

It has also been shown in preliminary analyses that 5 sessions of Default Mode Network-targeted cTBS improves processing speed in people with schizophrenia and substance use (t(9)=3.311, p=.009). This provides 1) reassuring evidence that Default Mode Network-targeted cTBS will not worsen cognitive performance; and 2) further support for our scientific hypotheses that Default Mode Network-targeted cTBS may improve cognitive performance.

These data show that Default Mode Network-targeted cTBS corrects abnormal DMN connectivity and reduces craving in SZ, supporting our hypothesis that Default Mode Network-targeted cTBS will normalize DMN connectivity and reduce cannabis craving.

Brief rTMS Treatments Can Safely Test the Effectiveness of Longer Treatment in the Future. In addition to its effectiveness as a treatment, rTMS is also a versatile research tool whose stimulation parameters can be changed. Depending on the parameters, rTMS can be excitatory or inhibitory. Intermittent theta burst stimulation (iTBS) and continuous theta burst stimulation (cTBS) are types of rTMS. iTBS is associated with excitatory effects which increase connectivity, while cTBS is associated with inhibitory effects which decrease connectivity. rTMS is FDA-approved for smoking cessation and can change brain network connectivity and craving in many substance use disorders.

Existing studies of rTMS for cannabis use in control and schizophrenia samples have targeted the dorsolateral prefrontal cortex (DLPFC) with modest effects on craving and use. These mixed findings suggest that perhaps DLPFC is not the ideal rTMS target for schizophrenia and that the parietal DMN might be more effective.

In this study, 2 rTMS interventions will be compared in a crossover design: 1) 5 sessions of rTMS delivered to the Default Mode Network (as previously have performed in schizophrenia) and 2) 5 sessions of rTMS delivered to the L DLPFC (as in FDA-approved treatment for major depressive disorder). The researchers will test if a 5-session rTMS intervention can cause short-term changes in 1) resting-state network functional connectivity, 2) cue-induced craving, and 3) cognitive performance in both healthy individuals who use cannabis and people with schizophrenia or schizoaffective disorder who use cannabis. The researchers here test a model that integrates brain network pathophysiology and cognition to 1) explain the extremely high prevalence of cannabis use in schizophrenia and 2) identify a treatment target for future clinical trials in schizophrenia and schizoaffective disorder.

Previous studies by our group and others have demonstrated the ability of rTMS to change patterns of activity in cortical networks of the human brain. In addition, the research team has also previously demonstrated the ability to both increase and decrease connectivity within a specific network (e.g. DMN) by neuroanatomically targeted rTMS. In the present study, one rTMS intervention will be delivered to the parietal node of the DMN, a region linked to cannabis use in schizophrenia in a network key to attentional and working memory performance, and one rTMS intervention will be delivered to the L DLPFC, a region responsible for executive function, an aspect of cognition key to reducing substance use. When previously applied a single session of rTMS to a parietal node of the DMN in individuals with schizophrenia, it was observed a significant effect on craving.

ELIGIBILITY:
Inclusion Criteria for Psychosis Participants:

* Age between 18-65 years
* Diagnosis of a psychotic disorder according to DSM-5 criteria and confirmed by SCID Current cannabis use (confirmed by urine cannabis testing)
* Must be able to read, speak and understand English
* Must be judged by study staff to be capable of completing the study procedures
* Participants will be in stable outpatient psychiatric treatment and psychiatrically stable with no recent (within the past 30 days) psychiatric hospitalizations or changes in their psychiatric medication regimens.

Inclusion Criteria for Healthy Controls:

- All of the above except for participants will not have a diagnosis of a psychotic disorder nor a first-degree relative with a psychotic disorder.

Exclusion Criteria for ALL participants:

* DSM-5 intellectual disability
* Substance use disorder (other than cannabis or nicotine) within the past three months
* Positive urine drug screen for illicit substance use that can increase seizure risk (cocaine, benzodiazepines, amphetamine, methamphetamine)
* Any history of a progressive or genetic neurologic disorder (e.g. Parkinson's disease, multiple sclerosis, tuberous sclerosis, Alzheimer's Disease) or acquired neurological disease (e.g. stroke, traumatic brain injury, tumor), including intracranial lesions
* History of head trauma resulting in any loss of consciousness (>15 minutes) or neurological sequelae
* Current history of poorly controlled headaches including chronic medication for migraine prevention
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* Any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g. MRI compatible joint replacement)
* Any devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt unless cleared by the responsible covering MD
* All female participants of child-bearing age will be required to have a pregnancy test; any participant who is pregnant or planning to become pregnant will not be enrolled in the study
* Medications will be reviewed by the responsible covering physician and a decision about inclusion will be made based on the participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and use of CNS active drugs. The published TMS guidelines review of medications to be considered with rTMS will be taken into consideration given their described effects on cortical excitability measures.
* Any changes in medications or hospitalizations within the past 30 days.
* Participants who, in the investigator's opinion, might not be suitable for the study or would be unable to tolerate the study visit

These exclusion criteria strictly follow all recommended guidelines as endorsed by the International Federation of Clinical Neurophysiology and the International Society for Transcranial Stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Efficacy: Determine if rTMS affects cue-induced craving and if craving change correlates with change in functional connectivity (n=100). | Up to 12 weeks
  Cue-induced craving will be measured using a 0-10 Visual Analog Scale (VAS) before, during, and after in-scanner presentation of visual cannabis cues. Whole DMN and L DLPFC-left insula connectivity will be calculated.

SECONDARY OUTCOMES:
2. Resting-state functional connectivity | Up to 12 weeks.
  The investigators will evaluate the effect of DMN-targeted cTBS on functional connectivity of the left parietal node of the DMN and the entire default mode network. The investigators will also evaluate the effect of L DLPFC-targeted iTBS on functional connectivity of the L DLPFC.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Reasonable requests for data will be considered.